CLINICAL TRIAL: NCT03488173
Title: Pharmacokinetic Study of Lansoprazole Capsules in Healthy Chinese Volunteer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Collaborators: Beijing Xuze Medical Technology Co., LTD. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: LC00-018-01
Record Dates: First submitted 2018-03-20; First posted 2018-04-04 (Actual); Last update posted 2019-08-15 (Actual); Status verified 2019-07

CONDITIONS: Effect of Drugs; Safety Issues
MeSH Terms: interventions — Lansoprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lansoprazole Capsules (Experimental): Lansoprazole Capsules 30 mg of Beijing Sihuan Pharm
  Interventions: Drug: Lansoprazole capsules
- Lansoprazole enteric-coated Capsules (Active Comparator): Lansoprazole enteric-coated Capsules 30 mg of Takeda Pharmaceutical Company Limited
  Interventions: Drug: Lansoprazole capsules

INTERVENTIONS:
Drug: Lansoprazole capsules — Test 1: 30 healthy volunteers will be included and randomized into 3 groups (10 for each). During the study session, subjects will receive a single dose of Lansoprazole capsules 30 mg in sequence of T-R-R in group A; R-T-R in group B; and R-R-T in group C.
  Test 2: 12 healthy volunteers will be recruited and randomized to 2 groups (6 for each). Subjects in group A will receive a single dose of experimental drug in sequence of fast-fed condition; while in group B, subjects will receive the same dose and drug but in fed-fast order.

SUMMARY:
The objective of this study was to compare pharmacokinetic of Lansoprazole Capsules 30 mg with Lansoprazole Capsules of Takeda 30 mg in healthy adult human subjects.

DETAILED DESCRIPTION:
i. randomized, open label, single-dose, two-treatment, three-period,partial replicate pharmacokinetic study of Lansoprazole 30 mg Capsules of Beijing Sihuan Pharm, comparing with that of Lansoprazole enteric-coated Capsules 30 mg of Takeda Pharmaceutical Company Limited in healthy, adult, human subjects under fasting conditions.

ii. randomized, open label, single dose, two-period, pharmacokinetic study of Lansoprazole 30 mg Capsules of Beijing Sihuan Pharm in healthy, adult, human subjects under fasting/fed conditions.

ELIGIBILITY:
Inclusion Criteria:

* Subject who were healthy, adult, human beings within 18 and 60 years of age (both inclusive)
* Male (weight ≥50kg) or female (weight ≥45kg); Subject having a body mass index between 19.0 and 26.0 (both inclusive), calculated as weight in Kg/height in m2.
* Subject who totally understand the aim, procedure, benefits and adverse effects of this clinical trial, make decision by his/her free will, and sign a consent form to follow the progress;
* The participant could communicate well with investigator, comply with and finish the study according to the procedure.

Exclusion Criteria:

* Subject who has past or present history of any serious diseases, including (but not limited to) digestive, cardiovascular, respiratory, urinary, musculoskeletal, endocrine, psychiatric or neurological, hematologic, immunological or metabolic disorders;
* Allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator;
* Intake of over the counter (OTC) or prescribed medications or vitamins or any traditional medicine products for the last 14 days before first dosing.
* Has a special requirement for food and cannot adhere to a uniform diet or swallowing victims.
* Venous puncture intolerable and/or blood phobia
* Abused of tea, coffee and caffeine-contained beverages; or taking caffeine/xanthene containing food or beverages (like tea, coffee, chocolates and cola drinks) for the last 48 hrs before first dosing.
* Habit of alcoholism; or frequent drinkers for the last 6 months before screening; or intake of any alcoholic products for the last 24 hrs before first dosing.
* Regular smoker who has a habit of smoking more than five cigarettes per day for the last 3 months and has difficulty in abstaining from smoking during sample collection period.
* Blood donation or blood loss ≥ 450 mL for the last 3 months before first dosing; or plan to donate blood or blood composition during the study or 3 months after the end of the study.
* Intake of any enzyme modifying food or beverages for the last 48 hrs before first dosing.
* Female detected to be pregnant, breast feeding or who is likely to become pregnant during the study; or subjects declined to practice non-pharmacologic prevention of birth control during the study.
* Abused of drugs or Intake of drugs for the last 3 months before screening.
* Subjects who had participated in any other clinical investigation using experimental drug/medical instrument/diagnostic reagent in past 3 months before screening.
* Clinically significant abnormalities judged by investigators during screening test.
* Confirmed positive in alcohol screening, smoking screening or selected drug of abuse.
* Human immunodeficiency virus(HIV), hepatitis B virus (HBV), hepatitis C virus (HCV) or syphilis positive.
* Other reasons for non-inclusion judged by investigator.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2018-04-23 (Actual); Primary Completion 2018-07-19 (Actual); Study Completion 2019-04-24 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics Assessment | 16 hrs post-dose on day 1.
  1. Cmax: Maximum Observed Plasma Concentration for lansoprazole Maximum observed plasma concentration (Cmax) is the peak plasma concentration of a drug after administration, obtained directly from the plasma concentration-time curve.
     [Time Frame: 16 hours post-dose on Day 1]
  2. TmaxTime to Reach the Maximum Plasma Concentration [Time Frame: 16 hours post-dose on Day 1]
  3. AUC(0-inf): Area Under the Plasma Concentration-time Curve from Time 0 to Infinity for lansoprazole AUC (0-inf) is a measure of total plasma exposure to the drug from time zero extrapolated to infinity [Time Frame: Time Frame: 16 hours post-dose on Day 1]
  4. AUC(0-16h): Area Under the Plasma Concentration-Time Curve From Time 0 to 36 hours Postdose for lansoprazoleAUC(0-36h) is measure of area under the plasma concentration and time curve from Time 0 to 36 hours postdose.
  [Time Frame: 16 hours post-dose on Day 1] model.

CONTACTS AND LOCATIONS:
Overall Officials: Lihua Wu, Doctor, Principal Investigator — First Affiliated Hospital of Zhejiang University; Jian Liu, Master, Principal Investigator — First Affiliated Hospital of Zhejiang University
Locations (1):
- First affiliated hospital of Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No